CLINICAL TRIAL: NCT01749891
Title: A Safety And Efficacy Study Of ALG-1001 In Human Subjects With Wet Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allegro Ophthalmics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Focus 3
Record Dates: First submitted 2012-12-06; First posted 2012-12-17 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Macular Degeneration
Keywords: Age Related Wet Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — risuteganib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1.5 mg ALG - 1001 (Experimental): Arm 1.5 mg ALG- 1001 per 50ul
  Interventions: Drug: ALG 1001
- Arm 2.5 mg ALG -1001 (Experimental): Arm 2.5 mg ALG -1001 per 50ul
  Interventions: Drug: ALG 1001
- Arm 4.0 mg ALG -1001 (Experimental): Arm 3 4.0 mg ALG -1001 per 50ul
  Interventions: Drug: ALG 1001

INTERVENTIONS:
Drug: ALG 1001 — Patients who will receive three, monthly intravitreal injections of 1.5mg, 2.5mg ,or 4.0 /50μl of ALG-1001 in 0.05cc in isotonic saline solution.
  Other Names: ALG-1001

SUMMARY:
The general objective of this study is to evaluate the safety and efficacy of ophthalmic intravitreal injections of ALG-1001 in human subjects with wet age-related macular degeneration (Wet AMD). This study builds upon the safety and efficacy results of numerous animal studies and an earlier Phase I Human Study in end-stage diabetic macular edema patients.

DETAILED DESCRIPTION:
The general objective of this study is to evaluate the safety and efficacy of ophthalmic intravitreal injections of ALG-1001 in human subjects with wet age-related macular degeneration (Wet AMD). This study builds upon the safety and efficacy results of numerous animal studies and an earlier Phase I Human Study in end-stage diabetic macular edema patients.

The specific objective of this six-month study is to evaluate the safety and efficacy of three monthly ophthalmic intravitreal injections of ALG-1001 in human subjects with Wet AMD, and to follow these subjects for an additional four months off-treatment. Three cohorts have been established as part of the study design, utilizing three different doses.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 50 years of age or older.
2. Active wet macular degeneration (AMD).
3. Subfoveal CNV (choroidal neovascular membrane) secondary to AMD in the study eye less than or equal to 12 MPS disc areas.
4. CNV greater than 50% of lesion area.
5. CNV may be classic, minimally classic, or occult.
6. For minimally classic and occult lesions in the study eye, must demonstrate decrease in BCVA (best corrected visual acuity) that must be assessed based on clinical exploration, macular thickening, presence of subretinal fluid or hemorrhage, and/or OCT findings consistent with CNV.
7. Study eye has a BCVA of 20/50 to 20/320 ETDRS (Early Treatment Diabetic Retinopathy Study )equivalent (65 letters to 23 letters), which in the opinion of the investigator is primarily due to Wet AMD.
8. Decrease in BCVA must be assessed based on clinical exploration, macular thickening, and/or fluorescein angiography consistent with CNV.
9. Intra-Ocular Pressure (IOP) is under control, IOP ≤ 25 mm.
10. Willing and able to return for all study visits.
11. Able to meet the extensive post-op evaluation regimen.
12. Patient can understand and sign informed consent form.
13. If subject is a female less than 60 years old, negative pregnancy test during the screening window.

Exclusion Criteria:

1. Media opacities or abnormalities that would preclude observation of the retina.
2. Other retinal pathologies that would interfere with the patient's vision.
3. Presence of other causes of CNV, including pathologic myopia, OHS (ocular histoplasmosis syndrome), angioid streaks, choroidal rupture or multifocal choroiditis in the study eye.
4. RPE (retinal pigment epithelium) rip or tear in the study eye.
5. Patients with current or prior retinal detachments, retinal tears, or tractional detachments in either eye.
6. A history of cataract surgery complications/vitreous loss in the study eye.
7. A history of penetrating ocular trauma in the study eye.
8. Chronic or recurrent uveitis.
9. Has undergone a vitrectomy (anterior or pars plana) in the study eye.
10. Ongoing ocular infection or inflammation in either eye.
11. A history of intravitreal injections of any type in the study eye within the last 45 days prior to study enrollment.
12. A history of cataract surgery complications/vitreous loss in the study eye.
13. Congenital malformations in the study eye.
14. Mentally handicapped.
15. Pregnant or a nursing female.
16. Currently participating in any other clinical research study
17. Contraindication to the study medication.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06-04 (Actual); Study Completion 2013-06-07 (Actual)

PRIMARY OUTCOMES:
Observation of dose limiting toxicity. | 6 months
  The primary endpoint of this study is observation of dose limiting toxicity and the maximum tolerated dose. The determination will be made by ocular adverse events by standard clinical ophthalmic evaluation, visual acuity changes at baseline by slit lamp biomicroscopy, tonometry, indirect ophthalmoscopy/ fundus photography, fluorescein angiography, OCT (optical coherence tomography) central macular thickness.

SECONDARY OUTCOMES:
Changes in OCT central macular thickness | 6 months
  Changes in OCT Central Macular Thickness

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Guerrero-Narranjo, MD, Principal Investigator — APEC Hospital Mexico City
Locations (1):
- APEC Hospital La Ceguera, Mexico City, Mexico